CLINICAL TRIAL: NCT03760250
Title: Open-label, Single-arm Pilot Study of the Effects of Topical 5% Imiquimod Cream on Preventing Keloid Recurrence After Surgical Keloidectomy
Brief Title: Imiquimod for Preventing Keloid Recurrence
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Investigator decision
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Thomas Leung M.D., Ph.D., Assistant Professor of Dermatology, University of Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 831625
Record Dates: First submitted 2018-11-28; First posted 2018-11-30 (Actual); Results first posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Keloid
MeSH Terms: conditions — Keloid | interventions — Imiquimod

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Imiquimod (Experimental): 5% Imiquimod cream once daily to keloid area 5-times a week for 6 weeks, starting 1-week prior to keloid excision
  Interventions: Drug: Imiquimod 5% cream

INTERVENTIONS:
Drug: Imiquimod 5% cream — Imiquimod 5% Cream application to keloid skin area 5-times per week for 6 weeks, starting 1-week before keloid excision
  Other Names: Aldara

SUMMARY:
This is an open-label, single-arm, pilot study on the effects of topical imiquimod treatment in preventing keloid recurrence after surgical excision. Keloids are abnormal scars that form in certain genetically predisposed individuals following trauma to the skin. They can be physically disabling and cause social impairment. Many therapies have been proposed and trialed for the permanent removal of keloids, but they all have limited efficacy. Topical imiquimod therapy has been reported to decrease keloid recurrence following keloidectomy in human patients. Given all previous reports of adjuvant imiquimod therapy to keloidectomy initiated imiquimod therapy after keloidectomy, the investigators would like to test the efficacy of topical imiquimod pre-treatment in preventing keloid recurrence after surgical excision. Therefore, the investigators are initiating an open-label pilot study of 10 patients age 18 or greater with keloids on the trunk and extremities excluding the groin and hands and feet who present to the dermatology clinic for standard of care keloid excision. Key exclusion criteria include vulnerable populations, immunocompromised state, hypersensitivity to study drug components, and keloids outside of specified areas. The main study intervention will be 6 weeks of treatment with topical 5% imiquimod cream, starting 1 week prior to surgical excision.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or greater
* Men and women who present clinically with keloids requesting excision
* Any number of keloids
* Keloid no larger than 5cm in diameter at the base
* Clinical findings consistent with keloid formation
* Location of keloid in low-risk areas - areas other than above the neck, hands, feet, or groin
* Able and willing to give informed consent

Exclusion Criteria:

* Age < 18
* Hypersensitivity to Imiquimod or to any of the excipients (methylhydroxybenzoate, propylhydroxybenzoate, cetyl alcohol, and stearyl alcohol)
* Involvement in a trial of another experimental intervention within 30 days
* Life threatening disease
* Use of immunosuppressive medications such as oral corticosteroids
* Bleeding disorders
* Not available for follow-up for 10 weeks
* Pregnant, intention to become pregnant during treatment phase of trial, or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-02-05 (Actual); Primary Completion 2019-09-05 (Actual); Study Completion 2020-09-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Imiquimod
Started | 6
Completed | 4
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Imiquimod
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Keloid Recurrence
Description: To assess the efficacy of 5% Imiquimod cream on decreasing keloid recurrence after excision when initiated prior to excision
Time Frame: 12 weeks after surgical excision
Measure: Count of Participants; unit: Participants
Arm/Group | Imiquimod
Number analyzed (Participants) | 4
Participants
  Recurred | 3
  Did not recur | 1

2. Secondary Outcome: Tolerability - Local Site Reaction Rated on a Scale
Description: tolerability of 5% imiquimod cream - clinical evaluation of local site reactions by clinicians for symptoms such as redness, discomfort, swelling, and ulceration at the site of drug application on the following scale with none being the best and severe the worst: none (no reaction in application site), mild (slight redness in application site), moderate (redness with swelling and pain in application site), severe (redness, swelling, ulceration in application site)
Time Frame: 12 weeks after surgical excision
Measure: Count of Participants; unit: Participants
Arm/Group | Imiquimod
Number analyzed (Participants) | 4
Participants
  local site reaction: none | 0
  local site reaction: mild | 4
  local site reaction: moderate | 0
  local site reaction: severe | 0

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Imiquimod
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2019-03-18): https://cdn.clinicaltrials.gov/large-docs/50/NCT03760250/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2019-03-15): https://cdn.clinicaltrials.gov/large-docs/50/NCT03760250/Prot_SAP_001.pdf